CLINICAL TRIAL: NCT07301476
Title: Evaluation of Local Anesthetic Diffusion to the Sciatic Nerve During Adductor Canal Block: an Observational Study
Brief Title: Evaluation of Local Anesthetic Diffusion to the Sciatic Nerve During Adductor Canal Block
Acronym: DiffuCAdd
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250730; 2025-A00945-44 (Registry Identifier: IDRCB)
Record Dates: First submitted 2025-11-18; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Sciatic Nerve; Adductor Canal Syndrome
Keywords: Adductor Canal; Sciatic Nerve; Local anesthesia diffusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adductor canal block is an effective analgesic technique for major knee surgery. However, the saphenous nerve block is not sufficient to explain this block's efficiency. It has been shown that adductor canal block can spread to the tibial and fibular nerves through the adductor hiatus. However, this diffusion's frequency has never been measured. The main objective of this study is to assess clinically the frequency of the spread of the adductor canal block to the fibular and tibial nerves.

DETAILED DESCRIPTION:
Adductor canal block is an effective analgesic technique for major knee surgery. The PROSPECT group recommends this block in first intention for locoregional anesthesia in total knee arthroplasty. It has been shown to not be inferior to femoral nerve block in this indication.

The adductor canal block targets the saphenous nerve and, through its spread in the adductor canal, the posterior branch of obturator nerve and the vastus medialis nerve. However, these nerves can't fully explain this block's efficiency.

It has been shown that local anesthetic can spread in the adductor canal to the tibial and fibular nerves through the adductor hiatus. However, this spread is inconstant, and no study has evaluated the frequency of this spread yet.

The main objective of this study is to assess the diffusion's frequency of adductor canal block to fibular and tibial nerves through clinical sensorimotor testing.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old scheduled for elective knee surgery under general anesthesia
* in our center
* receiving an adductor canal block

Exclusion Criteria:

* patients cognitively impaired,
* patients suffering from peripheral neuropathy at the lower limb,
* patients receiving an IPACK block or surgical knee infiltration to complete the adductor canal block analgesia.
* patients who refused to take part in this study
* pregnant or breastfeeding patients
* patients under guardianship
* imprisoned patients,
* patients without any medical insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be all the consecutive patients scheduled for elective knee surgery under general anesthesia in our center and receiving an adductor canal block.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of local anesthetic's spread to tibial and fibular nerve | at 4 hours
  The primary outcome is the frequency of local anesthetic's spread to tibial and fibular nerve during an adductor canal block, assessed by sensory and motor testing of these nerve territories.
  Sensorimotor testing will be performed at four hours with loco-regional anaesthesia.

SECONDARY OUTCOMES:
Frequency of reduction of sensitivity to cold or touch or reduction in MRC score | at 1 hour and at 4 hours
  Frequency of reduction of sensitivity to cold or touch or reduction in MRC score in fibular and tibial nerves territories assessed at one and four hours after the adductor canal block has been performed, as well as reduction of sensitivity to cold or touch in saphenous nerve territory assessed at one and four hours after nerve block.
Spread of the local anesthetic in the popliteal fossa | at baseline
  Qualitative assessment of local anaesthetic spread in the popliteal fossa on ultrasound recording (spread or no spread).
Evaluation of the positive and negative predictive value | at baseline and 1 hour, 4 hours
  Evaluation of the positive and negative predictive value, sensitivity and specificity, and positive and negative likelihood ratio of ultrasound-visualised diffusion to the tibial and fibular nerves as a predictive test for clinical impairment of the sensitivity and motor function of these nerves at 1 hour or 4 hours
Clinical alteration assessement | at Baseline and at 1 hour and 4 hours
  Clinical alteration of sensibility and motricity will be assessed before the adductor canal block is performed and then at H1 and H4. The ultrasound scan of the popliteal fossa will be performed at the same time as the local anaesthetic is administered.

CONTACTS AND LOCATIONS:
Overall Officials: Romuald Henry, MD, Principal Investigator — CHU Raymond Poincaré - APHP
Locations (1):
- Department of Anesthésia, CHU Raymond Poincaré - APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No